CLINICAL TRIAL: NCT04560036
Title: Hypoxia Measurement With FAZA PET/MRI in Patients With Metastasized Gastro-Oesophageal Cancer
Brief Title: FAZA PETMRI Gastro-Oesophageal Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 19-5849
Record Dates: First submitted 2020-09-11; First posted 2020-09-23 (Actual); Last update posted 2025-03-30 (Actual); Status verified 2025-03

CONDITIONS: Metastasized Gastro-Oesophageal Cancer

STUDY DESIGN:
Intervention Model Description: FAZA PET/MRI scan
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- FAZA PET/MRI scan (Other): FAZA PET/MRI scan before and after the standard of care chemotherapy
  Interventions: Diagnostic Test: FAZA PET/MRI scan

INTERVENTIONS:
Diagnostic Test: FAZA PET/MRI scan — FAZA PET/MRI scan before and after the standard of care chemotherapy

SUMMARY:
This is a single arm, pilot study of PET/MRI scan with radiotracer 18F-Fluoroazomycin Arabinoside (FAZA) before and after standard of care platinum-based chemotherapy for patients with metastasized Gastro-Oesophageal Cancer.

Gastroesophageal cancer (GEC) accounted for 2,3000 deaths in Canada in 2017 and majority of the patients present or develop metastatic disease following diagnosis. These patients are treated with platinum-based chemotherapy. There is currently no biomarker that can be used to predict the therapy responses. Additionally, patients that do not respond to the chemotherapy often deteriorate rapidly and are unable to receive second line therapy. Intratumoral hypoxia (low oxygen concentration) is a signature feature of aggressive and resistant tumour phenotype. Accurately predicting hypoxia in solid tumours offers an innovative and rational pradigm for predicting therapy responses. PET/MRI is an imaging technique combining the Positron Emission Tomography (PET) scan with Magnetic Resonance Imaging (MRI) scan. A radiotracer called 18F-Fluoroazomycin Arabinoside (FAZA) is used as a type of "dye" in the PET/MRI scan.

The primary goal of the study is to validate FAZA PET/MRI as a biomarker of hyupoxia in setting of gastro-oesophageal carcinoma. Patients with GEC will undergo FAZA PET/MRI scan before and after the standard of care chemotherapy. This would be correlated with clinical outcome in patients with metastatic GEC that have different responses to chemotherapy. Ultimately, we hope that the use FAZA PET/MRI in the study can help select the most effective treatment method for advanced GEC to extend life and improve quality of life while minimizing toxicity and healthcare costs.

The study subjects' clinical management will not be changed based on the PET-MR scan within the trial.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 years
* Patients with de novo or secondary metastasized gastro-oesophagesal cancer (adenocarcinoma)
* Glomerular Filtration rate> 45 ml/min
* No allergy to contrast agents

Exclusion Criteria:

* Contraindication for MR as per current institutional guidelines
* Inability to lie supine for at least 30 minutes
* Any patient who is pregnant or breastfeeding
* Any patient unable or unwilling to provide informed consent
* Patients who are allergic to ethanol as the FAZA preparation contains ethanol

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40 (Estimated)
Dates: Start 2020-09-15 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Validation of FAZA PET/MRI as a biomarker of hypoxia | two weeks before chemotherapy
  The FAZA uptake during the first PET/MRI scan
Validation of FAZA PET/MRI as a biomarker of hypoxia | 3 months after the chemotherapy
  The FAZA uptake during the 2nd PET/MRI scan

SECONDARY OUTCOMES:
Evaluate tumour marker ctDNA in blood samples | two weeks before chemotherapy
  Evaluate tumour marker ctDNA in blood samples
Evaluate tumour marker ctDNA in blood samples | 6 weeks after initiation of chemotherapy
  Evaluate tumour marker ctDNA in blood samples
Evaluate tumour marker ctDNA in blood samples | 3 months after chemotheray
  Evaluate tumour marker ctDNA in blood samples

CONTACTS AND LOCATIONS:
Overall Officials: Patrick Veit-Haibach, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- Univeristy Health Network, Toronto, Ontario, Canada